CLINICAL TRIAL: NCT03892317
Title: A Pharmacist Led, Patient Tailored Intervention to Improve Immunosuppressant Medication Adherence in Nonadherent Kidney Transplant Patients
Brief Title: Improving Adherence in Nonadherent Kidney Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 17HH4287
Record Dates: First submitted 2018-10-05; First posted 2019-03-27 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-10

CONDITIONS: Medication Adherence; Kidney Transplantation
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medication adherence interventions (Other): Pharmacist led medication adherence interventions which will be tailored to individual patient need
  Interventions: Behavioral: Pharmacist led medication adherence interventions

INTERVENTIONS:
Behavioral: Pharmacist led medication adherence interventions — Medication adherence interventions which will be tailored to individual patient need

SUMMARY:
Organs for transplantation remain a scarce and precious resource with over 5000 patients currently on the kidney transplant waiting list. A kidney transplant costs approximately £17,000 in the first year and £5,000 per subsequent year. If the transplant fails, the patient must return to dialysis at an estimated cost of £30,800 per year or be retransplanted. While short term outcomes have improved steadily over the last 15-20 years, longer term outcomes haven't and after 10 years approximately 30% of kidney transplants have failed. Nonadherence to immunosuppressive medication is increasingly being associated with these poor long term outcomes and studies have estimated that 30- 50% of transplant patients are nonadherent to their immunosuppressive medication. The investigators want to determine whether immunosuppression medication adherence can be improved in a group of patients receiving tailored medication adherence support form a pharmacist. Adherence support will be provided for one year and will be individualised to each patient in the intervention group after identifying both their practical and perceptual barriers to adherence. The adherence interventions offered may include additional education and medication counselling, setting alarms, provision of a medication list, the use of a medications adherence app on a smart phone, reducing the number and frequency of tablets a patient takes or referral on to another health professional such as a social worker or psychologist for additional support. A range of clinical outcomes will be assessed for all patients on a regular basis in order to determine whether the provision of effective medication adherence support for the kidney transplant patients may help to optimise the long-term outcomes of these transplants

DETAILED DESCRIPTION:
This study will be undertaken using a prospective, multidimensional design. 42 nonadherent kidney transplant patients will be included in the intervention group. The nonadherent patients will be identified through Imperial College Renal and Transplant Centre (ICRTC) Outpatient Clinic based at Hammersmith Hospital. Standard and transplant specific demographics will be collected for all patients. All kidney transplant patients have their tacrolimus levels measured at each clinic visit. The variability of these levels can be used as a marker of their adherence. Patients with a high intrapatient variability (IPV) of their levels are said to be nonadherent. The Chief Investigator or another member of the research team will approach individual patients directly in the transplant out-patient clinic where they are members of the multidisciplinary clinical care team. The Chief Investigator or another member of the research team may also telephone patients to invite them to clinic to discuss participation in the trial. The Chief Investigator or another member of the research team will describe the study to the patient, answer any questions they have and provide them with a participant information sheet (PIS). Patients will be given the opportunity to take the PIS away and think about whether they would like to participate. A follow up discussion either in clinic or on the phone will be arranged with the patient to answer any queries they have within two weeks of providing them with the PIS; during that discussion, the Chief Investigator or other member of the research team will arrange an appointment in the transplant clinic with the patient to sign the consent form if they do decide to participate. Patients recruited into the study will receive pharmacist led, patient tailored interventions to improve immunosuppressant medication adherence. Patients will be included in the study for one year from recruitment.

The pharmacist led, patient tailored intervention will involve regular, intensive, personalised support from a pharmacist to improve adherence to immunosuppressive medications. The pharmacist will meet with the patient on a regular basis in the transplant clinic to identify their perceptual and practical barriers to adherence and agree a support plan that is tailored to them.

Within the first two weeks of recruitment, the study pharmacist will meet with the patient in transplant clinic to:

* Undertake a full medication history
* Discuss self-reported medication nonadherence
* Undertake the BAASIS questionnaire
* Ask the patient to complete a Beliefs about Medicines Questionnaire (BMQ)
* Undertake a socioeconomic and educational assessment
* Undertake to gain collateral reporting of nonadherence by clinicians, relatives, friends or carers
* Perform a tacrolimus pill count
* Check in-house dispensing records of tacrolimus
* Identify barriers to adherence
* Tailor interventions and support to the needs of the patient
* Complete a motivational interview
* Agree to meet again during an outpatient clinic visit within an agreed time which is appropriate for the patient needs and within 3 months.

This first visit will provide a baseline assessment of the patient's medication adherence.

Tailored support may include:

* Setting alarms
* Medication diary card or calendar
* Medication compliance aid filled by the patient, family/carers or by a pharmacy professional
* Adherence app
* Reducing the complexity of the medication regime
* Positioning medication within their daily routine eg. by toothbrush
* Changing formulations
* Additional education regarding need for medication / timing of doses
* Referral to a social worker to assist with affordability of medicines
* Referral to a psychologist to explore deeper psychological issues regarding medicines taking

The structure of each follow up adherence review will be the same as the first formal adherence review with the exception that the BMQ will only be repeated at the end of the one year follow-up and the socioeconomic and educational assessment will only be undertaken at the first assessment review. Every patient will have a formal adherence assessment at recruitment and then at 3, 6, 9 and 12 months. At the end of one year of follow-up, the specific benefits perceived by the patient of intensive adherence support from a pharmacist will be determined through a questionnaire.

Baseline nonadherence will be measured at the first visit with the study pharmacist within two weeks of recruitment and then at 3, 6, 9 and 12 months. The IPV of their tacrolimus levels and their outpatient clinic nonattendance rate will be measured retrospectively in the 12 months prior to recruitment to the study and then prospectively at the end of the intervention year. The IPV is calculated from the tacrolimus levels measured for an individual patient using the coefficient of variance mathematical formula - Coefficient of variance (COV) defined as: SD x 100 / Mean. The outpatient clinic nonattendance for each participant will be taken from the hospital integrated computer system.

ELIGIBILITY:
Inclusion Criteria:

* Adult kidney transplant patients (18 years of age and above)
* Kidney transplant patients with an IPV of tacrolimus levels of greater than 18.15% in the previous 12 months

Exclusion Criteria:

* Antibody incompatible transplants including patients with preformed HLA and blood group incompatible
* Previous rejection
* Donor specific antibody positive
* HIV positive patients
* Simultaneous pancreas and kidney patients
* Paediatric patients (less than 18 years of age)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Goodall, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- Imperial College Renal and Transplant Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Bleser L, Matteson M, Dobbels F, Russell C, De Geest S. Interventions to improve medication-adherence after transplantation: a systematic review. Transpl Int. 2009 Aug;22(8):780-97. doi: 10.1111/j.1432-2277.2009.00881.x. Epub 2009 Apr 6. PMID 19386076
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Transplant Work Group. KDIGO clinical practice guideline for the care of kidney transplant recipients. Am J Transplant. 2009 Nov;9 Suppl 3:S1-155. doi: 10.1111/j.1600-6143.2009.02834.x. PMID 19845597
- [Background] Denhaerynck K, Steiger J, Bock A, Schafer-Keller P, Kofer S, Thannberger N, De Geest S. Prevalence and risk factors of non-adherence with immunosuppressive medication in kidney transplant patients. Am J Transplant. 2007 Jan;7(1):108-16. doi: 10.1111/j.1600-6143.2006.01611.x. Epub 2006 Nov 15. PMID 17109727
- [Background] Fine RN, Becker Y, De Geest S, Eisen H, Ettenger R, Evans R, Rudow DL, McKay D, Neu A, Nevins T, Reyes J, Wray J, Dobbels F. Nonadherence consensus conference summary report. Am J Transplant. 2009 Jan;9(1):35-41. doi: 10.1111/j.1600-6143.2008.02495.x. PMID 19133930
- [Background] Gaston RS, Hudson SL, Ward M, Jones P, Macon R. Late renal allograft loss: noncompliance masquerading as chronic rejection. Transplant Proc. 1999 Jun;31(4A):21S-23S. doi: 10.1016/s0041-1345(99)00118-9. No abstract available. PMID 10372038
- [Background] Morrissey PE, Flynn ML, Lin S. Medication noncompliance and its implications in transplant recipients. Drugs. 2007;67(10):1463-81. doi: 10.2165/00003495-200767100-00007. PMID 17600393
- [Background] Morrissey PE, Reinert S, Yango A, Gautam A, Monaco A, Gohh R. Factors contributing to acute rejection in renal transplantation: the role of noncompliance. Transplant Proc. 2005 Jun;37(5):2044-7. doi: 10.1016/j.transproceed.2005.03.017. PMID 15964334
- [Background] Prendergast MB, Gaston RS. Optimizing medication adherence: an ongoing opportunity to improve outcomes after kidney transplantation. Clin J Am Soc Nephrol. 2010 Jul;5(7):1305-11. doi: 10.2215/CJN.07241009. Epub 2010 May 6. PMID 20448067
- [Background] Schafer-Keller P, Steiger J, Bock A, Denhaerynck K, De Geest S. Diagnostic accuracy of measurement methods to assess non-adherence to immunosuppressive drugs in kidney transplant recipients. Am J Transplant. 2008 Mar;8(3):616-26. doi: 10.1111/j.1600-6143.2007.02127.x. PMID 18294158
- [Background] Wiebe C, Nevins TE, Robiner WN, Thomas W, Matas AJ, Nickerson PW. The Synergistic Effect of Class II HLA Epitope-Mismatch and Nonadherence on Acute Rejection and Graft Survival. Am J Transplant. 2015 Aug;15(8):2197-202. doi: 10.1111/ajt.13341. Epub 2015 Jun 11. PMID 26095765
- [Background] Sellares J, de Freitas DG, Mengel M, Reeve J, Einecke G, Sis B, Hidalgo LG, Famulski K, Matas A, Halloran PF. Understanding the causes of kidney transplant failure: the dominant role of antibody-mediated rejection and nonadherence. Am J Transplant. 2012 Feb;12(2):388-99. doi: 10.1111/j.1600-6143.2011.03840.x. Epub 2011 Nov 14. PMID 22081892
- [Background] Roberts DM, Jiang SH, Chadban SJ. The treatment of acute antibody-mediated rejection in kidney transplant recipients-a systematic review. Transplantation. 2012 Oct 27;94(8):775-83. doi: 10.1097/TP.0b013e31825d1587. PMID 23032865
- [Background] Wiebe C, Gibson IW, Blydt-Hansen TD, Karpinski M, Ho J, Storsley LJ, Goldberg A, Birk PE, Rush DN, Nickerson PW. Evolution and clinical pathologic correlations of de novo donor-specific HLA antibody post kidney transplant. Am J Transplant. 2012 May;12(5):1157-67. doi: 10.1111/j.1600-6143.2012.04013.x. Epub 2012 Mar 19. PMID 22429309
- [Background] Pinsky BW, Takemoto SK, Lentine KL, Burroughs TE, Schnitzler MA, Salvalaggio PR. Transplant outcomes and economic costs associated with patient noncompliance to immunosuppression. Am J Transplant. 2009 Nov;9(11):2597-606. doi: 10.1111/j.1600-6143.2009.02798.x. PMID 19843035
- [Background] Butler JA, Roderick P, Mullee M, Mason JC, Peveler RC. Frequency and impact of nonadherence to immunosuppressants after renal transplantation: a systematic review. Transplantation. 2004 Mar 15;77(5):769-76. doi: 10.1097/01.tp.0000110408.83054.88. PMID 15021846
- [Background] Massey EK, Tielen M, Laging M, Timman R, Beck DK, Khemai R, van Gelder T, Weimar W. Discrepancies between beliefs and behavior: a prospective study into immunosuppressive medication adherence after kidney transplantation. Transplantation. 2015 Feb;99(2):375-80. doi: 10.1097/TP.0000000000000608. PMID 25606787
- [Background] Massey EK, Tielen M, Laging M, Beck DK, Khemai R, van Gelder T, Weimar W. The role of goal cognitions, illness perceptions and treatment beliefs in self-reported adherence after kidney transplantation: a cohort study. J Psychosom Res. 2013 Sep;75(3):229-34. doi: 10.1016/j.jpsychores.2013.07.006. Epub 2013 Aug 3. PMID 23972411
- [Background] Dew MA, DiMartini AF, De Vito Dabbs A, Myaskovsky L, Steel J, Unruh M, Switzer GE, Zomak R, Kormos RL, Greenhouse JB. Rates and risk factors for nonadherence to the medical regimen after adult solid organ transplantation. Transplantation. 2007 Apr 15;83(7):858-73. doi: 10.1097/01.tp.0000258599.65257.a6. PMID 17460556

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Medication Adherence Interventions
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Medication Adherence Interventions
Number analyzed (Participants) | 42
Age, Customized [Mean (Full Range); unit: years]
  Age at Transplant | 52.27 [43.89 to 60.65]
  Age at Recruitment | 58.45 [49.84 to 67.06]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 13
  Caucasian | 18
  Indoasian | 9
  Other | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 42
Marital Status [Count of Participants; unit: Participants]
  Cohabiting | 2
  Divorced | 4
  Married | 27
  Single | 7
  Widowed | 2
Education Status [Count of Participants; unit: Participants]
  A levels/B Tec | 11
  Degree | 11
  GCSE / O Levels | 12
  Higher Degree | 2
  No Qualification | 6
Graft Type [Count of Participants; unit: Participants]
  Living Donor | 22
  Deceased Donor | 20
Dialysis Modality [Count of Participants; unit: Participants]
  HD | 26
  PD | 2
  Pre-emptive | 14
Cause of ESRD [Count of Participants; unit: Participants]
  APKD | 6
  DM | 7
  GN | 12
  Other | 9
  Unknown | 6
  Urological | 2
Diabetes [Count of Participants; unit: Participants]
  Yes | 15
  No | 27

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Patients Being Adherent/Non-aherent After the Intervention
Description: Immunosuppression Medication adherence will be assessed and compared using the BAASIS questionnaire at recruitment and at the end of the study. The BAASIS questionnaire is a closed question questionnaire (either adherent or non-adherent); it is validated for assessing immunosuppression nonadherence in transplant patients. Any patient answering yes to any of the questions is assessed to be nonadherent
Time Frame: One year
Population: Any patient answering yes to any of the questions is assessed to be nonadherent. Results are reported at time 0 (baseline), time 3 months, time 6 months, time 9 months, and time 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Medication Adherence Interventions
Number analyzed (Participants) | 42
Participants
  Adherent (Time 0) | 15
  Adherent (Time 3 months) | 30
  Adherent (Time 6 months) | 34
  Adherent (Time 9 months) | 35
  Adherent (Time 12 months) | 36

2. Primary Outcome: Change in the Median IPV Before and After the Intervention
Description: Intrapatient variability of tacrolimus levels will be measured and compared and reported as percentage difference
Time Frame: One year
Measure: Mean (Full Range); unit: % difference
Arm/Group | Medication Adherence Interventions
Number analyzed (Participants) | 42
% difference | 32.03 [-22.61 to 80.83]

3. Primary Outcome: Change in Outpatient Clinic Nonattendance Rate Before and After the Intervention
Description: Data for this outcome measure has not been analysed: originally the outpatient clinic nonattendance rate was to be assessed and compared during the 12 months prior to recruitment to the study and during the study
Time Frame: One year
Population: Patients were not analysed for this outcome
Arm/Group | Medication Adherence Interventions
Number analyzed (Participants) | 0

4. Secondary Outcome: Biopsy Proven ACR / AMR
Description: Number of patients who develop biopsy proven ACR/AMR
Time Frame: One year
Population: No biopsies were indicated throughout the study
Measure: Count of Participants; unit: Participants
Arm/Group | Medication Adherence Interventions
Number analyzed (Participants) | 42
Participants | 0

5. Secondary Outcome: The Number of Readmissions
Description: The number of readmissions and their reasons why during the study will be recorded
Time Frame: One year
Population: Some patients who had readmissions had more than one readmission.
Measure: Count of Participants; unit: Participants
Arm/Group | Medication Adherence Interventions
Number analyzed (Participants) | 42
Participants
  Number of readmissions associated with the study | 0
  Number of patients who had readmissions | 12
  Number of patients who didn't have readmissions | 30

6. Secondary Outcome: Donor Specific Antibody (DSA) or Transplant Glomerulopathy
Description: For secondary outcome measures 6&7 - no one developed a Donor Specific Antibody (DSA) or Transplant Glomerulopathy, Fibrosis, Hyalinosis, Calcineurin Inhibitor (CNI) Toxicity or Diabetic Change.
  Number of patients who develop a DSA or transplant glomerulopathy (CNI) toxicity or diabetic change on biopsy
Time Frame: One year
Measure: Number; unit: number of interventions
Arm/Group | Medication Adherence Interventions
Number analyzed (Participants) | 42
number of interventions | 0

7. Secondary Outcome: Fibrosis, Hyalinosis, Calcineurin Inhibitor (CNI) Toxicity or Diabetic Change on Toxicity
Description: For secondary outcome measures 6&7 - No biopsies were indicated throughout the study therefore no one developed Fibrosis, Hyalinosis, Calcineurin Inhibitor (CNI) Toxicity or Diabetic Change
  Number of patients who develop fibrosis, hyalinosis, calcineurin inhibitor
Time Frame: One year
Measure: Number; unit: number of interventions
Arm/Group | Medication Adherence Interventions
Number analyzed (Participants) | 42
number of interventions | 0

8. Secondary Outcome: Graft Loss
Description: Number of patients who lose their graft
Time Frame: One year
Measure: Count of Participants; unit: Participants
Arm/Group | Medication Adherence Interventions
Number analyzed (Participants) | 42
Participants | 0

9. Secondary Outcome: Death
Description: Number of patients who die
Time Frame: One year
Measure: Count of Participants; unit: Participants
Arm/Group | Medication Adherence Interventions
Number analyzed (Participants) | 42
Participants | 0

10. Secondary Outcome: Serum Creatinine
Description: Change in serum creatinine at the end of the study Data for this outcome measure has not been analysed
Time Frame: One year
Reporting Status: Not Posted

11. Secondary Outcome: eGFR
Description: Change in eGFR at the end of the study. Data for this outcome measure has not been analysed
Time Frame: One year
Reporting Status: Not Posted

12. Secondary Outcome: Proteinuria
Description: Change in proteinuria at the end of the study. Data for this outcome measure has not been analysed
Time Frame: One year
Reporting Status: Not Posted

13. Secondary Outcome: Haematocrit
Description: Change in haematocrit at the end of the study. Data for this outcome measure has not been analysed
Time Frame: One year
Reporting Status: Not Posted

14. Secondary Outcome: Haemoglobin
Description: Change in haemoglobin at the end of the study. Data for this outcome measure has not been analysed
Time Frame: One year
Reporting Status: Not Posted

15. Secondary Outcome: Albumin
Description: Change in albumin at the end of the study. Data for this outcome measure has not been analysed
Time Frame: One year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 yr circa
Description: There are no significant adverse events attributed to the study.
Arm/Group | Medication Adherence Interventions
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 14/42
Other Adverse Events (participants affected / at risk) | 38/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medication Adherence Interventions (N=42)
Infection - Tx kidney (Renal and urinary disorders) | 2 (2)
Infection - native kidney (Renal and urinary disorders) | 2 (2)
Infection - Tx gynae (Reproductive system and breast disorders) | 1 (1)
Infection - chest (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infection - colecystis (Gastrointestinal disorders) | 1 (1)
ITP (Vascular disorders) | 1 (1)
NODAT (Metabolism and nutrition disorders) | 1 (1)
Elective Surgery (Surgical and medical procedures) | 2 (2)
Pain - Ostheopatic fracture spine (Musculoskeletal and connective tissue disorders) | 1 (1)
Angioedema and hyponatraemia (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medication Adherence Interventions (N=42)
Infection - colecystitis (Renal and urinary disorders) | 1 (1)
Infection - EBV (Infections and infestations) | 1 (1)
Infection - COVID (loss of sense of taste and smell) (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pain - hip and knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - generalised aches and pains (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - hernia (Gastrointestinal disorders) | 1 (1)
Swollen hand - possible gout (General disorders) | 1 (1)
Fall (General disorders) | 1 (1)
NODAT - new diagnosis (Surgical and medical procedures) | 1 (1)
AKI and high tacrolimus levels post ibuprofen ingestion (General disorders) | 1 (1)
Kidney biopsy - no new changes (Surgical and medical procedures) | 1 (1)
Hypertensive (Vascular disorders) | 1 (1)
Thrombocytopenia in relation to ITP (Vascular disorders) | 1 (1)
BCC removal (Surgical and medical procedures) | 1 (1)
Bowens disease - new diagnosis (Skin and subcutaneous tissue disorders) | 1 (1)
Heamorrhagic cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Increased frequency of nightmares (General disorders) | 1 (1)
Colonoscopy to investigate iron deficiency anaemia (Surgical and medical procedures) | 1 (1)
OGD as pre-planned procedure (Surgical and medical procedures) | 1 (1)
Flexible cystoscopy - enlarged prostate (benign) (Renal and urinary disorders) | 1 (1)
Concern expressed by patient over memory decline (Psychiatric disorders) | 1 (1)
Worsening symptoms of established SVCO (Vascular disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Hypocalcaemia (Blood and lymphatic system disorders) | 1 (1)
Lump at site of flu vaccine (General disorders) | 1 (1)
Intermittent itch - resolved (General disorders) | 1 (1)
Hayfever (Immune system disorders) | 1 (1)
Loss of appetite (Metabolism and nutrition disorders) | 1 (1)
Hysteroscopic removal of IUD as an OP (Surgical and medical procedures) | 1 (1)
SAD (General disorders) | 1 (1)
Carotid endarterectomy as elective procedure - preplanned (Surgical and medical procedures) | 1 (1)
Intolerant of doxazosin (Immune system disorders) | 1 (1)
Cateract removal - preplanned (Surgical and medical procedures) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Keloid scar removal as OP daycase - longstanding (Surgical and medical procedures) | 1 (1)
Weight increase (Metabolism and nutrition disorders) | 1 (1)
Mouth ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Sclerosing mesenteritis (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/17/NCT03892317/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT03892317/ICF_001.pdf